CLINICAL TRIAL: NCT00529425
Title: Postoperative Analgesia With Local Infiltration After Femoral Neck Fracture vs. Traditional Treatment of Pain With Opioids
Brief Title: Postoperative Analgesia With Local Infiltration After Femoral Neck Fracture
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S-VF-20060072 - femoral neck
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Last update posted 2010-05-06 (Estimated); Status verified 2010-04

CONDITIONS: Femoral Neck Fracture
Keywords: Femoral neck fracture; Hip fracture
MeSH Terms: conditions — Femoral Neck Fractures; Hip Fractures | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ropivacaine (Active Comparator)
  Interventions: Drug: Ropivacaine
- Saline (Placebo Comparator)
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine

SUMMARY:
Reducing pain is an essential factor for early mobilization after osteosynthesis of femoral neck fractures. Systemic opioids have side effects that might obstruct mobilization and induce delirium and nausea. The investigators hypothesized that wound infiltration results in reduction in systemic opioid usage and pain relief without side effects.

ELIGIBILITY:
Inclusion Criteria:

* Femoral neck fracture
* Fracture due to low energy trauma
* Ability to understand danish and give informed consent
* Ability to walk before trauma
* Indication for osteosynthesis
* ≥ 8 in OMC (Orientation-Memory-Concentration) test with a possible maximum of 28 points
* Informed consent

Exclusion Criteria:

* Drug or medical abuse
* Drug intolerance
* Pathological fractures
* Inflammatory arthritis
* Patient included in the study with the contralateral hip

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-01; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Consumption of opioids

SECONDARY OUTCOMES:
Pain

CONTACTS AND LOCATIONS:
Overall Officials: Soren Overgaard, Professor, MD, DmSc, Study Chair — Odense University Hospital, DK-5000 Odense C, Denmark; Rune Dueholm Bech, MD, Principal Investigator — Odense University Hospital, DK-5000 Odense C, Denmark
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Bech RD, Lauritsen J, Ovesen O, Emmeluth C, Lindholm P, Overgaard S. Local anaesthetic wound infiltration after internal fixation of femoral neck fractures: a randomized, double-blind clinical trial in 33 patients. Hip Int. 2011 Mar-Apr;21(2):251-9. doi: 10.5301/HIP.2011.6513. Epub 2011 Apr 5. PMID 21484739